CLINICAL TRIAL: NCT01364415
Title: A Phase I, Multi-center, Open-label, Dose Escalation Study of Pasireotide (SOM230) LAR in Patients With Advanced Neuroendocrine Tumors (NETs)
Brief Title: Dose Escalation Study of Pasireotide (SOM230) in Patients With Advanced Neuroendocrine Tumors (NETs)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230D2101
Record Dates: First submitted 2011-05-18; First posted 2011-06-02 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-06

CONDITIONS: Neuroendocrine Tumors
Keywords: MTD; pasireotide; LAR; NETs; advanced neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pasireotide

ARMS (1):
- Pasireotide LAR (Experimental)
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide LAR
  Other Names: SOM230

SUMMARY:
This study designed to determine the Maximum Tolerated Dose (MTD) for patients with advanced Neuroendocrine Tumors (NETs) and to characterize the safety, tolerability, Pharmacokinetics and preliminary efficacy of pasireotide LAR administered i.m. once every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 yrs old, histologically confirmed advanced well or moderately differentiated neuroendocrine tumor/carcinoma
* unresectable metastatic NET tumor with measurable disease
* life expectancy ≥ 12 weeks

Exclusion Criteria:

* Patients with CNS metastases who are neurologically unstable or requiring increasing doses of steroids to control their CNS disease
* patients with known hypersensitivity to somatostatin analogs
* patients with symptomatic cholelithiasis in the past 2 months
* patients with history of another known primary malignancy with exception of non-melanoma skin cancer or carcinoma in situ of uterine cervix
* patients with known history of hepatitis C or chronic active hepatitis B
* patients with diagnosis of HIV.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determine the MTD/RP2D of pasireotide LAR when administered i.m. q28 days to patients with advanced NETs | Sequentiona 56 day cohorts until the MTD is determined
  Frequency of dose-limiting toxicities (DLTs) at each dose level associated with q28 days administration of pasireotide LAR during the first 2 treatment cycles.

SECONDARY OUTCOMES:
assess the safety and tolerability of pasireotide LAR | minimum of twelve 28 day cycles to approximately eighteen 28 day cycles
  Incidence of adverse drug events, overall and by severity and incidence of serious adverse events and laboratory abnormalities. Also, changes in laboratory assessments, electrocardiograms, Holter monitor, imaging for gallstones, and assessment of physical examinations such as vital signs
assess the pharmacokinetics (PK) of pasireotide LAR | minimum of twelve 28 day cycles to approximately eighteen 28 day cycles
  Pasireotide Cmax and Ctrough
assess the pharmacodynamics (PD) of pasireotide LAR | minimum of twelve 28 day cycles to approximately eighteen 28 day cycles
  Changes from baseline values in IGF-1, chromogranin A and neuron-specific enolase
assess the preliminary efficacy (anti-tumor activity) of pasireotide LAR. | minimum of twelve 28 day cycles to approximately eighteen 28 day cycles
  Disease control rate (CR+PR+SD as assessed by RECIST 1.0). Also measure progression free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center Cedars Sinai 4, Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Institute SC-1, Tampa, Florida
  - Dana Farber Cancer Institute SC-6, Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center UT MD Anderson Cancer Ctr, Houston, Texas

REFERENCES:
- [Derived] Yao JC, Chan JA, Mita AC, Kundu MG, Hermosillo Resendiz K, Hu K, Ravichandran S, Strosberg JR, Wolin EM. Phase I dose-escalation study of long-acting pasireotide in patients with neuroendocrine tumors. Onco Targets Ther. 2017 Jun 27;10:3177-3186. doi: 10.2147/OTT.S128547. eCollection 2017. PMID 28721067
- See also: Results for CSOM230D2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15767